CLINICAL TRIAL: NCT05216029
Title: Study of Efficacy of Oncology Dashboard in Improving Operational Efficiency and Patient Outcomes
Brief Title: Oncology Dashboard for the Improvement of Operational Efficiency and Patients Outcomes in Patients With Sarcoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-0707; NCI-2021-09453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0707 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (oncology dashboard) (Experimental): Radiologist records information from patient's recent scan into oncology dashboard. Patients view images of how disease may have changed over time on oncology dashboard.
  Interventions: Other: Informational Intervention; Other: Questionnaire Administration
- Group II (standard of care) (Experimental): Patients receive standard of care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Other: Informational Intervention — View oncology dashboard
  Arms: Group I (oncology dashboard)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial investigates whether measuring and presenting information about a patient's cancer treatment to them, their doctor, and their radiologist using a tool called an "oncology dashboard" may help patients understand the disease better and help the patient's medical team manage their care more efficiently. The oncology dashboard tool may help patients understand the disease better and may help improve the efficiency of their medical care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the changes in oncology workflow times from baseline to follow up visits between intervention (follow-up visit with oncology dashboard tool) and control (follow-up visit without oncology dashboard tool) groups.

SECONDARY OBJECTIVES:

I. To compare the changes in radiology workflow times from baseline to follow up visits between intervention (follow-up visit with oncology dashboard tool) and control (follow-up visit without oncology dashboard tool) groups.

II. Assess and compare the proportion of patients who correctly indicate the changes in tumor size while on therapy at the baseline and at the follow-up visit (with the oncology dashboard tool).

IIa. Compare the change in proportion of patients who correctly indicate the changes in tumor size while on therapy from baseline to follow-up visit between intervention and control groups.

III. Assess the patient's satisfaction with physician communication during the clinic visit and with the current treatment plan at each visit for each group.

IV. Assess changes in the radiology report quality with the following measures (all changes will be compared between intervention and control groups):

IVa. Whether or not the current study was compared to the imaging study that was performed at the start of current therapy.

IVb. The number of time points reviewed by the radiologist. IVc. The time interval between the earliest study reviewed and the current study.

IVd. Percentage of target lesions measured and listed in the radiology report. V. In patients who have stable disease or mildly progressive disease at the time of the baseline assessment, assess the impact of patient understand on the decision to continue and discontinue therapy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Radiologist records information from patient's recent scan into oncology dashboard. Patients view images of how disease may have changed over time on oncology dashboard.

GROUP II: Patients receive standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoma on active chemotherapy/targeted therapy
* Patients must have stable to mildly progressive disease or better on baseline assessment

  * Baseline measurement and follow-up measurement have to be performed on the same treatment for consistency. If patients with progressive disease are included into the study at baseline, follow-up measurement will be on a different treatment. Invariable, initiation of a new treatment, in the setting of progressive disease, lengthens oncology workflow which would affect the post measurement
* Patients must have been on the same treatment for at least 6 weeks
* Patients must have at least 3 prior imaging studies of the same body part/tracked lesion/area of interest separated by 6 weeks or more between studies
* Patients should be continuing same therapy for the next 6-8 weeks
* Patients must have plan for follow-up with imaging studies at MD Anderson Cancer Center (MDACC) while on therapy
* Patients who are receiving therapy outside of MDACC but having their follow-up imaging at MDACC are eligible
* >= 18 years of age

Exclusion Criteria:

* Expected survival of less than 8 weeks
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 4
* Non- English-speaking patients and patients with cognitive impairment who cannot complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Time to complete medical oncology review (oncology workflow) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Ravi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org